CLINICAL TRIAL: NCT05030272
Title: Comparing Two Behavioral Approaches to Quitting Smoking in Mental Health Settings
Acronym: MTQT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00110770; R01DA047301 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-07

CONDITIONS: Tobacco Use Disorder; Mental Illness; Recurring Major Depressive Disorder; Bipolar Disorder; Schizophrenia; Schizoaffective Disorder; Persistent Depressive Disorder
MeSH Terms: conditions — Tobacco Use Disorder; Mental Disorders; Bipolar Disorder; Schizophrenia; Psychotic Disorders | interventions — Crisis Intervention; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- "Quit on the Go" (formerly "Learn to Quit") (Experimental): A smartphone app developed by the research team designed for people with serious mental illness, that provides Acceptance and Commitment Therapy skills to address (a) smoking cessation and (b) mental health symptoms. This app intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches and a 5-10 week course of NRT gum (or Nicotine Lozenges if unable to use gum). Participants also receive technical smartphone coaching for the first 4 weeks of the study.
  Interventions: Device: Quit on the Go App (formerly "Learn to Quit " App); Drug: Nicotine patch; Behavioral: Smartphone coaching; Drug: Nicotine gum; Drug: Nicotine Lozenges
- Brief Advice (Standard of Care) (Other): Brief Advice and Combined Nicotine Replacement Therapy (patches and gum or lozenges) has been recommended by the US Clinical Practice Guidelines for patients with psychiatric illness. Brief Advice will consist of 20 minutes of guidance about the use of nicotine replacement therapy, and strategies to initiate and maintain a quit attempt. The intervention is combined with an 8-week course of nicotine replacement therapy (NRT) patches and a 5-10 week course of NRT gum (or Nicotine Lozenges if unable to use gum).
  Interventions: Behavioral: Brief advice; Drug: Nicotine patch; Drug: Nicotine gum; Drug: Nicotine Lozenges

INTERVENTIONS:
Device: Quit on the Go App (formerly "Learn to Quit " App) — A smartphone app developed by the research team designed for people with serious mental illness, that provides Acceptance and Commitment Therapy skills to address (a) smoking cessation and (b) mental health symptoms.
  Arms: "Quit on the Go" (formerly "Learn to Quit")
Behavioral: Brief advice — Brief Advice will consist of 20 minutes of guidance about the use of nicotine replacement therapy, and strategies to initiate and maintain a quit attempt.
  Arms: Brief Advice (Standard of Care)
Drug: Nicotine patch — All participants will receive an 8-week course of transdermal nicotine patches. The first 4 weeks of use will be 21mg/24 hours, followed by 2 weeks of 14mg/24 hours patches, and finally 2 weeks of 7mg/24 hours patches.
  Other Names: NRT
Behavioral: Smartphone coaching — Participants randomized to the smartphone app intervention will receive 4 weeks of smartphone coaching given by research staff. The coaching is meant to be a time to address any issues that may rise with the participants' study smartphone or app.
  Arms: "Quit on the Go" (formerly "Learn to Quit")
Drug: Nicotine gum — Each participant enrolled will be given NRT gum (5-10week course) to be taken orally as nicotine cravings arise. Depending on participants' nicotine dependence, they will receive either the 2mg or 4mg (if they smoke within the first 30 minutes of waking) gum pieces per package instructions. We will direct subjects to use them for the first weeks following their quit date, using no more than one every 1-2 hours.
  Other Names: NRT
Drug: Nicotine Lozenges — In cases where participants are unable to chew nicotine gum, lozenges will be sent as a replacement of Nicotine gum. Depending on participants' nicotine dependence, they will receive either the 2mg or 4mg (if they smoke within the first 30 minutes of waking) lozenge pieces per package instructions. We will direct subjects to use them for the first weeks following their quit date, using no more than one every 1-2 hours.
  Other Names: NRT

SUMMARY:
The study team will conduct a Multisite Randomized Controlled Trial to evaluate the advantages and disadvantages of two approaches for quitting smoking among people with serious mental illness (SMI). The study will compare a novel app tailored to people with SMI, Quit on the Go, to a standard of care smoking cessation intervention. We will test the effectiveness of the Quit on the Go app, an intervention that has demonstrated feasibility and acceptability in the target population, as a tool for smoking cessation in people with SMI. Participants with SMI will be recruited across 3 sites (Duke University, Univ. at Buffalo, and Wake Forest University).

DETAILED DESCRIPTION:
Smoking tobacco shortens the lifespan of adults with serious mental illness by 25 years and contributes to 317 billion dollar expenditures in healthcare, indirect loss of earnings and disability benefits. Determining whether it is possible to deliver more effective and wider reaching smoking cessation interventions to individuals with serious mental illness is a high priority. Smartphone apps are a wide-reaching technology that could provide individuals with serious mental illness the necessary skills for quitting. However, our research has shown that apps developed for the general public have inadequate levels usability and engagement in people with serious mental illness.

In a previous pilot trial of a tailored smoking cessation app for people with serious mental illness, Learn to Quit (NCT03069482), we identified successful recruitment and retention methods for smokers with SMI, demonstrated a 4-fold increase in objectively measured interactions of the novel app, obtained promising cessation rates for the experimental app (12% for Quit on the Go formerly "Learn to Quit" versus 3% for NCI QuitGuide), and identified a reliable methodological approach to conduct a fully-powered randomized controlled trial.

Based on this pilot work, we plan to conduct a clinical trial to test this new model in a diverse and representative sample of the SMI population. Specifically, the proposed trial will test whether a tailored smoking cessation app for people with serious mental illness, Quit on the Go, results in higher levels of smoking abstinence compared to a standard of care intervention for this psychiatric population, Brief Advice. Both interventions will receive combined nicotine replacement therapy. The second aim of this trial is to test a mechanistic model of app efficacy by examining mediators of app engagement and treatment outcomes. Finally, the trial will evaluate the cost-effectiveness of these interventions to inform public health policy regard the use of mHealth in this population.

In a multi-site, two-arm randomized controlled trial, 450 individuals with serious mental illness will be randomly assigned to one of two conditions. In the experimental condition, participants will use the Quit on the Go app. In the comparator condition, participants will receive Brief Advice for smoking cessation. Participants in both conditions will receive combined Nicotine Replacement Therapy (standard dosing of nicotine patch plus 5 week course of nicotine gums). Study duration will be 6 months, with 3 follow-up appointments at 1-month, 3-month, and 6-months. Our proposed methods are appropriate given our established procedures during our pilot trial regard to participant assignment, delivery of interventions, data collection and analysis (NCT03069482).

The proposed study meets NIDA's major programmatic priorities of using innovative technologies (e.g., smartphones) and integrating behavioral and pharmacological interventions to improve substance use treatment and outcomes (NOT-DA-10-019). The proposal addresses a serious problem -- high smoking rates in people with SMI -- in a high priority, high cost population, by delivering a novel behavioral intervention for smoking cessation in "real-world" settings. If shown to be effective, the proposed intervention will provide a new model for delivering inexpensive, widely accessible smoking cessation interventions in adults with SMI.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of schizophrenia, schizoaffective, bipolar, recurring major depressive disorder or Persistent Depressive Disorder
2. Functional impairment as indicated by a score of 2 or greater on the WHODAS 8 item version
3. Smoker as indicated by smoking greater than or equal to 5 cigarettes per day over the past 6 months;
4. Desire to quit smoking as indicated by self-reported serious intention to quitting tobacco within the next 6 months;
5. Age 18 and older;
6. Willing and medically eligible to use NRT;
7. Currently receiving psychiatric treatment and intent to receive treatment for the duration of the study (therapy, medications, etc.).

Exclusion Criteria

1. Problematic substance use, as defined by the Addiction Severity Index, within the last 30 days, twice within the past 6 months, or hospitalization for substance abuse within the past year.
2. Current acute psychotic episode or unsafe to participate in the study as defined by the Mini International Neuropsychiatric Interview for Psychotic Disorders (Sheehan et al., 1998);
3. Being pregnant or the intention to become pregnant in the next 6 months;
4. Currently receiving any pharmacological and/or behavioral intervention or counseling for smoking cessation;
5. Currently using e-cigarettes or other tobacco products besides cigarettes > 10 days in the past 30 days.
6. Unsafe to participate in the study due to moderate or high risk of suicide determined by the Columbia-Suicide Severity Rating Scale (C-SSRS) - Screen Version, defined as answering 'yes' to both question 3 for the last month and 'yes' to question 6 for lifetime (moderate risk), or 'yes' to questions 4 and 5 for the recent month, or 'yes' to question 6 for the last 3 months (high risk).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
CO-verified 7-day point-prevalence abstinence at 6-month follow-up | 6 month follow-up
  Abstinence is determined by a self-report of not smoking any tobacco product for greater than or equal to 7 days prior to Week 24 and biochemically verified by an expired carbon monoxide breath test reading of < 5 ppm at Week 24. If the participant does not meet both criteria, they are not considered abstinent.
  As per convention, participants are assumed to be smoking if they report smoking at the time-point, cannot be reached to provide data at the time-point, fail to provide a breath sample at the time-point, or provide a breath sample at the time-point that is greater than or equal to 5 ppm.

SECONDARY OUTCOMES:
Change in average number of cigarettes smoked per day | 1 month follow-up
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Change in average number of cigarettes smoked per day | 3 month follow-up
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Change in average number of cigarettes smoked per day | 6 month follow-up
  Change in self-reported number of cigarettes smoked per day, averaged within groups.
Average number of quit attempts per group | 1 month follow-up
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking at all for 24 hours or more.
Average number of quit attempts per group | 3 month follow-up
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking at all for 24 hours or more.
Average number of quit attempts per group | 6 month follow-up
  Average number of quit attempts self-reported per group at the specified time point. Quit attempts are defined by no smoking at all for 24 hours or more.
Time to 7-day relapse | 1 month follow-up
  Average number of days of abstinence before relapse per group. Relapse defined by an instance of 7 consecutive days of smoking.
Time to 7-day relapse | 3 month follow-up
  Average number of days of abstinence before relapse per group. Relapse defined by an instance of 7 consecutive days of smoking.
Time to 7-day relapse | 6 month follow-up
  Average number of days of abstinence before relapse per group. Relapse defined by an instance of 7 consecutive days of smoking.
30-day point prevalence abstinence rates | 1 month follow-up
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days but < 30 days prior to the timepoint.
Biochemically confirmed 30-day point prevalence abstinence rates | 3 month follow-up
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days but < 30 days prior to the time point. Abstinence is determined by a self-report of not smoking any tobacco product at all during the corresponding time frame period, AND by a result of less than 5 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent.
Biochemically confirmed 30-day point prevalence abstinence rates | 6 month follow-up
  Percent of subjects in each group self-reporting no smoking at all for greater or equal to 30 days but < 30 days prior to the time point. Abstinence is determined by a self-report of not smoking any tobacco product at all during the corresponding time frame period, AND by a result of less than 5 ppm in carbon monoxide breath testing. If the participant does not meet both criteria, they are not considered abstinent.
Prolonged abstinence rates | 1 month follow-up
  Percent of subjects in each group reporting prolonged abstinence. Abstinence is determined by a self-report of not relapsing after their quit date (i.e., not smoking for 7 consecutive days, or not smoking at least once each week for 2 consecutive weeks) following a 2-week grace period.
Prolonged abstinence rates | 3 month follow-up
  Percent of subjects in each group reporting prolonged abstinence. Abstinence is determined by a self-report of not relapsing after their quit date (i.e., not smoking for 7 consecutive days, or not smoking at least once each week for 2 consecutive weeks) following a 2-week grace period.
Prolonged abstinence rates | 6 month follow-up
  Percent of subjects in each group reporting prolonged abstinence. Abstinence is determined by a self-report of not relapsing after their quit date (i.e., not smoking for 7 consecutive days, or not smoking at least once each week for 2 consecutive weeks) following a 2-week grace period.
Continuous abstinence rates | 1 month follow-up
  Percent of subjects in each group self-reporting continuous abstinence (no smoking at all) between target quit date and specified time point.
Continuous abstinence rates | 3 month follow-up
  Percent of subjects in each group self-reporting continuous abstinence (no smoking at all) between target quit date and specified time point. Biochemically verified (CO < 5 ppm).
Continuous abstinence rates | 6 month follow-up
  Percent of subjects in each group self-reporting continuous abstinence (no smoking at all) between target quit date and specified time point. Biochemically verified (CO < 5 ppm).

OTHER OUTCOMES:
Average app usability scores | 1 month follow-up
  Average self-reported scores of usability on the 10-item System Usability Scale. Scores range from 0-100 with higher scores indicating higher usability of the app.
Average user experience scores | 1 month follow-up
  Average self-reported scores of user experience using an adapted 5-item app user experience scale.
Average user experience scores | 3 month follow-up
  Average self-reported scores of user experience using an adapted 5-item app user experience scale.
Average user experience scores | 6 month follow-up
  Average self-reported scores of user experience using an adapted 5-item app user experience scale.
Average frequency of app use | Weeks 0-24
  Average frequency of app use over the 24-week study period. Measured by average number of app openings.
Average duration of app use | Weeks 0-24
  Average duration of app use over the 24-week study period.
Average number of app modules completed | Weeks 0-24
  Average number of app modules completed over the 24-week study period.
Average acceptance of physical smoking cravings | 1 month follow-up
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Average acceptance of physical smoking cravings | 3 month follow-up
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Average acceptance of physical smoking cravings | 6 month follow-up
  Average self-reported scores of acceptance of cravings on the physical sensations subscale of the Avoidance and Inflexibility Scale. Scores range from 4-20 with lower scores indicating more acceptance of smoking cravings.
Nicotine patch use | 3 month follow-up
  Average number of days (out of 56 possible) per arm that participants used the nicotine patch.
Nicotine gum use | 3 month follow-up
  Average number of nicotine gum used per arm.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vilardaga, PhD, Principal Investigator — Wake Forest University
Locations (3):
- United States (3):
  - University at Buffalo, Buffalo, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No